CLINICAL TRIAL: NCT05223998
Title: Manual Implantation of Full-Thickness Skin Microcolumns for 'Donor-Free' Skin Renewal
Brief Title: Manual Implantation of Full-Thickness Skin Microcolumns
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Metis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00071475; CDMRP-MB200033 (Other Grant/Funding Number: Congressionally Directed Medical Research Program Office)
Record Dates: First submitted 2021-10-20; First posted 2022-02-04 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Wound of Skin; Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Intervention Model Description: Proof of concept
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Full-thickness skin microcolumns Implantation (Experimental): implantation of FTSM on open wound
  Interventions: Procedure: Full-thickness skin microcolumns implantation

INTERVENTIONS:
Procedure: Full-thickness skin microcolumns implantation — Surgical harvest and implantation of FTSM on an open wound requiring coverage.

SUMMARY:
The objective of this study is to validate the proof of concept regarding the approach of manual implantation of full-thickness skin microcolumns (FTSMs) as coverage for open wounds without creating an additional donor scar and while also capitalizing on the wound healing benefits offered by full-thickness skin grafts.

DETAILED DESCRIPTION:
Previously three patients have been successfully treated with the use of manual FTSM for wound coverage. To provide additional proof of concept data, this study will validate manual FTSM implantation on a larger scale with a 10-patient population. This will be measured by the following hypothesized parameters: time to re-epithelization, pigmentation, wound contraction, scar thickness, pain at the donor site and injury site healing outcome. The approach to testing this hypothesis will be to perform manual FTSM harvest, placement on the injured site, covered by an inert dressing for 10 patients with open wounds necessitating tissue coverage. The rationale is that although preliminary proof of concept data has already been obtained from three patients treated with FTSM implantation, additional proof of concept data would strengthen the conclusions made based on these cases.

ELIGIBILITY:
Inclusion Criteria:

* 8-85 years of age
* 10-125 cm2 open wound on the scalp, neck, torso or extremities necessitating tissue coverage
* Sufficiently healthy skin to serve as a donor site

Exclusion Criteria:

* Wound area involving the face*
* Wound area involving joints*
* Pregnancy
* Prisoner
* Active wound infection at potential treatment sites
* Exposed muscle, joint, tendon, or bone within the wound bed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11-04 (Estimated); Primary Completion 2025-09-29 (Estimated); Study Completion 2025-09-29 (Estimated)

PRIMARY OUTCOMES:
Donor site re-epithelization between day 10 to 14 | 10-14 days
  Donor site re-epithelization between day 10 to 14

SECONDARY OUTCOMES:
Donor site | up to 6 months
  Assess donor site pigmentation, contraction, scar thickness and pain
Injured site | up to 6 months
  Assess injured site re-epithelization, pigmentation, contraction, scar thickness and pain

CONTACTS AND LOCATIONS:
Overall Officials: Rodney Chan, MD, Principal Investigator — Metis Foundation

IPD SHARING:
Plan to Share IPD: No